CLINICAL TRIAL: NCT04887506
Title: Phase 3 Study Investigating the Efficacy and Safety of TAVT-45 (Abiraterone Acetate) Granules for Oral Suspension (Novel Abiraterone Acetate Formulation) Relative to a Reference Abiraterone Acetate Formulation in Patients With mCSPC & mCRPC
Brief Title: TAVT-45 (Abiraterone Acetate) Granules in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tavanta Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAVT45C02; 2020-005611-46 (EudraCT Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-14 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Metastatic Castration-sensitive Prostate Cancer; Metastatic Prostate Cancer
Keywords: Prostate; Metastatic; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAVT-45 (Experimental): TAVT-45 administered twice daily as a 1 x sachet containing TAVT-45 (250 mg abiraterone acetate) + Prednisone (5mg once or twice daily, depending on prostate cancer population). TAVT-45 administered approximately every 12 hours without respect to food. Patients treated for 84 days.
  Interventions: Drug: TAVT-45; Drug: Prednisone
- Reference abiraterone acetate (Zytiga®) - R-AA (Active Comparator): Zytiga (reference abiraterone acetate formulation, hereafter referred to as R-AA) administered once daily as (2 x 500mg Zytiga tablets) + Prednisone (5mg once or twice daily, depending on prostate cancer population). R-AA administered once daily either ≥ 1 hour before or ≥ 2 hours after a meal. Patients treated for 84 days.
  Interventions: Drug: Zytiga; Drug: Prednisone

INTERVENTIONS:
Drug: TAVT-45 — 250 mg abiraterone acetate granules for oral suspension in a sachet, reconstituted in water or specified fruit juice (orange juice), administered twice daily.
  Arms: TAVT-45
Drug: Zytiga — 500 mg tablet, two tablets administered once daily
  Other Names: Abiraterone Acetate
  Arms: Reference abiraterone acetate (Zytiga®) - R-AA
Drug: Prednisone — mCSPC patients received 5 mg orally once daily. mCRPC patients received 5 mg orally twice daily.
  Other Names: Encorton

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of a new formulation of an existing drug product called TAVT-45 in patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, open-label study to evaluate the pharmacodynamic effect and safety profile of TAVT-45 compared to Zytiga (reference abiraterone acetate formulation, hereafter referred to as R-AA) in patients with high-risk metastatic castrate sensitive prostate cancer (mCSPC) and metastatic castrate resistant prostate cancer (mCRPC). Randomization was stratified by prostate cancer population (CSPC vs CRPC) and baseline testosterone (<10 vs ≥ 10 ng/dL). Patients were treated for 84 days and randomized into one of two groups in a 1:1 ratio:

* TAVT-45: Administered twice daily as 1 x sachet containing TAVT-45 (250 mg abiraterone acetate), reconstituted in water or specified fruit juice (orange juice), + Prednisone (5 mg once or twice daily, depending on prostate cancer population)
* R-AA: Administered once daily as (2 x 500 mg Zytiga tablets) + Prednisone (5 mg once or twice daily, depending on prostate cancer population)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed
2. Male patients at least 18 years of age or older at time of consent
3. Pathologically confirmed adenocarcinoma of the prostate
4. Ongoing therapy with a gonadotropin releasing hormone (GnRH) agonist or antagonist (unless patient has already had a bilateral orchiectomy) AND serum testosterone level <50 ng/dL at screening
5. Have either metastatic CSPC or metastatic CRPC (per protocol definitions).
6. The following prior treatments and/or surgery for prostate cancer are allowed:

   1. CSPC:

      * Up to 90 days of androgen deprivation therapy (ADT) with gonadotropin-releasing hormone (GnRH) agonists/antagonists or orchiectomy with or without concurrent anti-androgens prior to patients' randomization is permitted
      * Patients may have one course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease (e.g., impending cord compression or obstructive symptoms) if administered prior to randomization
      * Radiation or surgical therapy that was not initiated 4 weeks after the start of ADT or orchiectomy
   2. CRPC:

      * Previous chemotherapy with docetaxel for metastatic disease with treatment completed at least 1 year prior to screening
7. Discontinuation of flutamide or nilutamide, and other anti-androgens prior to the start of study medication; discontinuation of bicalutamide prior to start of study medication
8. Discontinuation of strong cytochrome P450 3A4 (CYP3A4) inducers at least 4 weeks prior to start of study medication
9. Discontinuation of radiotherapy prior to start of study medication
10. Discontinuation of herbal supplements at least 4 weeks prior to the first dose of study medication and for the duration of the trial.
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at screening
12. Normal organ function with acceptable initial laboratory values within the screening period:

    * Absolute neutrophil count (ANC): ≥ 1,500/μl
    * Albumin: ≥ 3.0g/dL
    * Hemoglobin: ≥ 9g/dL
    * Platelet count: ≥ 100,000/μl
    * Serum Creatinine: ≤ 3.0 x the institutional upper limit of normal (ULN)
    * Potassium: ≥ 3.5 mmol/L (within institutional normal range)
    * Bilirubin: ≤ 1.5 ULN (unless documented Gilbert's disease)
    * Aspartate aminotransferase (AST): ≤ 2.5 x ULN
    * Alanine aminotransferase (ALT): ≤ 2.5 x ULN
13. Life expectancy of at least 6 months at screening
14. Patients engaged in sex with women of child-bearing potential agree to use a condom plus another effective contraception method. Patients agree to use a condom when engaged in any sexual activity, including sex with a pregnant woman. These restrictions will apply from the time informed consent is provided until 3 weeks after the last dose of study medication is taken.
15. Patient is willing and able to comply with all protocol requirements

Exclusion Criteria:

1. For mCSPC patients: any prior pharmacotherapy, radiation therapy, or surgery for metastatic prostate cancer not specified as allowable treatment in Inclusion Criterion 6. For example, prior therapy with apalutamide or enzalutamide is prohibited as well as therapy with an investigational agent as described in Exclusion Criterion 16.
2. For mCRPC patients:

   * Prior treatment with abiraterone or enzalutamide is prohibited
   * Previous chemotherapy is prohibited with exception of docetaxel treatment as specified in the inclusion criteria 6.
3. Initiation of bisphosphonate or denosumab therapy within 4 weeks prior to the start of study drug/reference product. Patients who are on a stable dose of these medications for at least 4 weeks at the time of starting study drug/reference product will be eligible.
4. Therapy with estrogen within 4 weeks prior to the start of study drug
5. Use of systemic glucocorticoids equivalent to >10 mg prednisone daily. Patients who have discontinued or reduced dosing to the equivalent of ≤ 10 mg prednisone daily within 14 days prior to the start of study drug are eligible
6. Known, symptomatic metastases to the brain or central nervous system involvement (patients with asymptomatic and neurologically stable disease for the past 4 weeks will be permitted)
7. History of adrenal gland dysfunction defined as requiring treatment for adrenal insufficiency
8. History of other malignancy within the previous 2 years (no longer being actively treated), with the exceptions of basal cell carcinoma, nonmuscle invasive bladder cancer that has been treated and is under surveillance, or other in-situ cancers with a low likelihood of recurrence
9. Major surgery within 4 weeks prior to the start of study drug
10. Known gastrointestinal disease or condition that could impair absorption inclusive of gastrocolic fistula, gastroenterostomy, biliary obstruction, cirrhosis, chronic pancreatitis or pancreatic cancer, cystic fibrosis, lactate deficiency, amyloidosis, celiac disease, Crohn's disease, radiation enteritis, intestinal resection, and history of bariatric surgery
11. Known history of human immunodeficiency virus or seropositive test for hepatitis C virus (HCV) or hepatitis B surface antigen (HBsAg) (note: HCV patients with undetectable viral load will be eligible)
12. Poorly controlled diabetes, defined as hemoglobin A1c (HbA1c) > 8% within the past 12 months
13. Uncontrolled hypertension at screening
14. History of New York Heart Association class III or IV heart failure
15. Serious concurrent illness, including psychiatric illness, that could interfere with study participation
16. Receipt of another investigational agent within 4 weeks or 5 x the treatment half-life, whichever is longer, of treatment start.
17. Known hypersensitivity or allergy to abiraterone acetate, prednisone or any excipients in the study drugs
18. In the opinion of the investigator, participation in the trial would prevent the patient from receiving local standard-of-care treatment for metastatic prostate cancer, if clinically indicated, after completion of the trial
19. Other condition which, in the opinion of the Investigator, would preclude participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Maetzel, MD, PhD, Study Chair — Tavanta Therapeutics inc.
Locations (40):
- United States (13):
  - Research Site, Homewood, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, San Bernardino, California
  - Research Site, Denver, Colorado
  - Research Site, Bradenton, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Jeffersonville, Indiana
  - Research Site, Annapolis, Maryland
  - Research Site, Troy, Michigan
  - Research Site, New York, New York
  - Research Site, Virginia Beach, Virginia
- France (2):
  - Research Site, Suresnes, Hauts-de-Seine
  - Research Site, Brest
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Debrecen
- Poland (5):
  - Research Site, Warsaw, Masovia
  - Research Site, Bydgoszcz
  - Research Site, Lublin
  - Research Site, Piaseczno
  - Research Site, Warsaw
- Research Site, Ponce, Puerto Rico
- Spain (9):
  - Research Site, Madrid, Arturo Soria, 270
  - Research Site, Madrid, Av. Reyes Católicos 2
  - Research Site, Manresa, Barcelona
  - Research Site, Madrid, Calle de Oña 10
  - Research Site, Barcelona, Sabadell
  - Research Site, Barcelona
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Seville
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Västerås
- United Kingdom (6):
  - Research Site, Torquay, Devon
  - Research Site, Cheltenham, Gloucestershire
  - Research Site, Hampstead, London
  - Research Site, Glasgow, Scotland
  - Research Site, Guildford, Surrey
  - Research Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsors website — https://www.tavanta.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 107 patients were randomized, and 103 patients received at least 1 dose of study medication (4 patients randomized to the R-AA arm were discontinued before receiving any study medication due to adverse event [n=1], lab result [n=1] and subject withdrawal [n=2]).
Groups:
- TAVT-45: TAVT-45 administered twice daily as a 1 x sachet containing TAVT-45 (250 mg abiraterone acetate) + Prednisone (5mg once or twice daily, depending on prostate cancer population). TAVT-45 administered approximately every 12 hours without respect to food. Patients treated for 84 days.
  TAVT-45: 250 mg abiraterone acetate granules for oral suspension in a sachet, administered twice daily.
  Prednisone: mCSPC patients received 5 mg orally once daily. mCRPC patients received 5 mg orally twice daily.
- Reference Abiraterone Acetate (Zytiga®) - R-AA: Zytiga (reference abiraterone acetate formulation, hereafter referred to as R-AA) administered once daily as (2 x 500mg Zytiga tablets) + Prednisone (5mg once or twice daily, depending on prostate cancer population). R-AA administered once daily either ≥ 1 hour before or ≥ 2 hours after a meal. Patients treated for 84 days.
  Zytiga: 500 mg tablet, administered twice daily.
  Prednisone: mCSPC patients received 5 mg orally once daily. mCRPC patients received 5 mg orally twice daily.
Period: Overall Study
Arm/Group | TAVT-45 | Reference Abiraterone Acetate (Zytiga®) - R-AA
Started | 54 | 53
Modified Intent-to-treat (mITT) Population (Modified intent-to-treat (mITT) population included all randomized patients who received at least one dose of study medication) | 54 | 49
Completed | 48 | 45
Not Completed | 6 | 8
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 4 | 3
Not completed — Other - Not Reported | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAVT-45 | Reference Abiraterone Acetate (Zytiga®) - R-AA | Total
Number analyzed (Participants) | 54 | 49 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 47 | 43 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (8.45) | 74.9 (8.40) | 74.7 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 49 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 50 | 45 | 95
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 51 | 44 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Poland | 5 | 2 | 7
  Spain | 19 | 19 | 38
  Sweden | 5 | 0 | 5
  United Kingdom | 10 | 6 | 16
  France | 2 | 2 | 4
  Hungary | 5 | 4 | 9
  United States | 8 | 16 | 24
Prostate Cancer Type [Number; unit: participants]
  metastatic castrate resistant prostate cancer (mCRPC) | 33 | 30 | 63
  metastatic castrate sensitive prostate cancer (mCSPC) | 21 | 19 | 40
Gleason score [Count of Participants; unit: Participants] — Gleason grading system refers to how abnormal the prostate cancer cells look via pathology and how likely the cancer is to advance and spread. A lower Gleason grade means that the cancer is slower growing and not aggressive.
  Participants
    Low (<7) | 3 | 7 | 10
    Medium (7) | 10 | 7 | 17
    High (8-10) | 38 | 35 | 73
    Missing | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Serum Testosterone (ng/dL) Days 9 and 10 Average (Rounded-up), CR-ITT
Description: The primary endpoint was the between group comparison of serum testosterone levels for the average of levels on Days 9 and 10 (rounded-up) for mCRPC patients.
Time Frame: Average over Day 9 and Day 10
Population: The mCRPC ITT (CR-ITT) population was a subset of the mITT population (all randomized patients who received at least one dose of study medication) and included mCRPC patients only.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/dL
Groups:
- TAVT-45 CR-ITT: All patients in the CR-ITT population treated with TAVT-45.
- R-AA CR-ITT: All patients in the CR-ITT population treated with R-AA.
Arm/Group | TAVT-45 CR-ITT | R-AA CR-ITT
Number analyzed (Participants) | 32 | 29
ng/dL | 1.0000 [1.000 to 1.000] | 1.0000 [1.000 to 1.000]
Statistical Analysis 1: Comparison: TAVT-45 CR-ITT vs R-AA CR-ITT; Primary analysis of equivalence of TAVT 45 and R AA based on average serum testosterone (ng/dL) (rounded up values of Days 9 and 10); Test type: Equivalence — If the 90% confidence interval (CI) fell within the recommended 0.800-1.250 limits of equivalence when analyzed on a natural log scale, then treatments were therapeutically equivalent based on rounded-up average Days 9 and 10 testosterone levels; Geometric mean ratio = 1 — The 90% CIs for the geometric mean ratio (GMR) were not evaluable

2. Secondary Outcome: Serum Testosterone (ng/dL) Days 9 and 10 Average (Rounded-up), CS-ITT
Description: This was a supplementary analysis of equivalence, with a between group comparison of serum testosterone for the Days 9 and10 average (rounded-up) values for mCSPC patients treated with either TAVT-45 or R-AA.
Time Frame: Average over Day 9 and Day 10
Population: The mCSPC ITT (CS-ITT) population was a subset of the mITT population and included mCSPC patients only.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/dL
Groups:
- TAVT-45 CS-ITT: All patients in the CS-ITT population treated with TAVT-45.
- R-AA CS-ITT: All patients in the CS-ITT population treated with R-AA.
Arm/Group | TAVT-45 CS-ITT | R-AA CS-ITT
Number analyzed (Participants) | 21 | 19
ng/dL | 1.01179 [0.98533 to 1.03896] | 1.03758 [1.00899 to 1.06697]
Statistical Analysis 1: Comparison: TAVT-45 CS-ITT vs R-AA CS-ITT; Supplementary analysis of equivalence of TAVT-45 and R-AA based on average serum testosterone (ng/dL) (rounded up values of Days 9 and 10) in the CS-ITT population; Test type: Equivalence — If the 90% CI fell within the recommended 0.800-1.250 limits of equivalence when analyzed on a natural log scale, then treatments were therapeutically equivalent based on rounded-up average Days 9 and 10 testosterone levels; Geometric mean ratio = 0.975, 90% CI 2-sided [0.944 to 1.007]

3. Secondary Outcome: Serum Testosterone (ng/dL) Days 9 and 10 Average (Rounded-up), mITT
Description: Supplementary analysis of equivalence of TAVT-45 and R-AA on Days 9 and 10 average (rounded-up) values in the mITT population (including mCRPC and mCSPC patients).
Time Frame: Average over Day 9 and Day 10
Population: mITT population: all randomized patients who received at least one dose of study medication.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/dL
Groups:
- TAVT-45 mITT: All patients in the mITT population treated with TAVT-45.
- R-AA mITT: All patients in the mITT population treated with R-AA.
Arm/Group | TAVT-45 mITT | R-AA mITT
Number analyzed (Participants) | 54 | 49
ng/dL | 1.00410 [0.99406 to 1.01425] | 1.01469 [1.00401 to 1.02548]
Statistical Analysis 1: Comparison: TAVT-45 mITT vs R-AA mITT; Supplementary analysis of equivalence of TAVT-45 and R-AA based on average serum testosterone (ng/dL) (rounded up values of Days 9 and 10) in the mITT population; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.99, 90% CI 2-sided [0.978 to 1.002]

4. Secondary Outcome: Percent of Subjects With PSA-50 Response, mITT
Description: The PSA-50 response is defined as a decrease of ≥ 50% in prostate-specific antigen (PSA) levels from baseline.
Time Frame: Response at any time over the 84-day post-treatment period.
Population: mITT population: all randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | TAVT-45 mITT | R-AA mITT
Number analyzed (Participants) | 54 | 49
Participants | 47 | 39
Statistical Analysis 1: Comparison: TAVT-45 mITT vs R-AA mITT; Test type: Equivalence — Odds ratio generated using the Wald method; p = 0.3408, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.574 to 4.979]

ADVERSE EVENTS:
Time Frame: From baseline to end of treatment (84 days)
Groups:
- TAVT-45: TAVT-45: 500 mg administered as 250 mg tablet twice daily (250 mg abiraterone acetate granules for oral suspension in a sachet, reconstituted in water or specified fruit juice [orange juice]) + Prednisone (5mg once or twice daily, depending on prostate cancer population).
  TAVT-45 administered approximately every 12 hours without respect to food. Patients treated for up to 84 days.
  Prednisone: mCSPC patients received 5 mg orally once daily. mCRPC patients received 5 mg orally twice daily.
- R-AA (Zytiga): R-AA: 1000 mg administered once daily as (2 x 500mg Zytiga tablets) + Prednisone (5mg once or twice daily, depending on prostate cancer population).
  R-AA administered either ≥ 1 hour before or ≥ 2 hours after a meal. Patients treated for up to 84 days.
  Prednisone: mCSPC patients received 5 mg orally once daily. mCRPC patients received 5 mg orally twice daily.
Arm/Group | TAVT-45 | R-AA (Zytiga)
All-Cause Mortality (participants affected / at risk) | 1/54 | 1/49
Serious Adverse Events (participants affected / at risk) | 5/54 | 3/49
Other Adverse Events (participants affected / at risk) | 38/54 | 36/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVT-45 (N=54) | R-AA (Zytiga) (N=49)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVT-45 (N=54) | R-AA (Zytiga) (N=49)
Alanine aminotransferase increased (Investigations) | 5 (6) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 3 (3)
Hypertension (Vascular disorders) | 9 (11) | 7 (10)
Hot flush (Vascular disorders) | 5 (5) | 2 (2)
Asthenia (General disorders) | 3 (3) | 4 (6)
Oedema peripheral (General disorders) | 2 (2) | 5 (5)
Fatigue (General disorders) | 3 (3) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
COVID-19 (Infections and infestations) | 6 (6) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT04887506/Prot_SAP_000.pdf